CLINICAL TRIAL: NCT05990010
Title: Prevalence of Obstructive Sleep Apnea Among Atrial Fibrillation Patients: A Cross-sectional Study From Jordan
Brief Title: OSA Prevalence in Atrial Fibrillation Patients: Jordanian Study
Status: Completed | Type: Observational
Sponsor: King Abdullah University Hospital (Other)
Responsible Party: Principal Investigator, Rashid Ibdah, Rashid Ibdah, MD, King Abdullah University Hospital
Other Study IDs: 22/130/2020
Record Dates: First submitted 2023-08-05; First posted 2023-08-14 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation; Obstructive Sleep Apnea
Keywords: AF; OSA; berlin questionnaire
MeSH Terms: conditions — Atrial Fibrillation; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with AF
  Interventions: Diagnostic Test: Berlin Questionnaire
- Patients without AF
  Interventions: Diagnostic Test: Berlin Questionnaire

INTERVENTIONS:
Diagnostic Test: Berlin Questionnaire — The Berlin Questionnaire is a simple survey that helps doctors identify OSA risk. It looks at snoring, daytime sleepiness, obesity, and hypertension. A positive score in two or more areas indicates high risk, while one or none suggests low risk. It is an easy and effective tool to assess OSA risk, with proven validity.

SUMMARY:
Current Knowledge:

Countless studies have been conducted to study the relationship between OSA and AF, and a significant association has been established between both diseases, owing to the numerous shared risk factors and a wide variety of pathophysiological changes resulting from both diseases being relevant to each other. Our study inspects this relationship from a cardiovascular standpoint, examining the prevalence of OSA in existing AF patients, which could be interpreted as AF being a risk factor for OSA development.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or above

Exclusion Criteria:

* Unable to give research consent
* Patients who were unwilling to complete the questionnaires
* Patients who suffer from mental illness

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who had visited King Abdullah University Hospital cardiology clinics within the timeframe of (2017-2019).
Sampling Method: Non-Probability Sample
Enrollment: 545 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
The Berlin Questionnaire survey | baseline
  Prevalence of Obstructive Sleep Apnea among Atrial Fibrillation Patients

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdullah University Hospital cardiology clinics, Irbid, Ramtha, Jordan

IPD SHARING:
Plan to Share IPD: Undecided